CLINICAL TRIAL: NCT01544517
Title: Five-day Concomitant Versus 10-day Sequential Therapy for Eradication of Helicobacter Pylori Infection: a Randomized Trial of Levofloxacin-based Regimens
Brief Title: 5 Day Concomitant Versus 10 Day Sequential Therapy for Eradication of H. Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco Romano, Associate Professor of Gastroenterology, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2010-02464415
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Concomitant therapy; Sequential therapy; levofloxacin
MeSH Terms: interventions — Amoxicillin; Esomeprazole; Tinidazole; Levofloxacin; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5d-QCT (Experimental): 5-day eradication regimen consisting in the concomitant administration of esomeprazole 40mg bid + amoxicillin 1g bid + levofloxacin 500mg bid + tinidazole 500mg bid
  Interventions: Drug: Eradication therapy (amoxicillin; esomeprazole; tinidazole; levofloxacin)
- 10-day sequential regimen (Active Comparator): 5 days of esomeprazole 40mg bid + amoxicillin 40mg bid followed by 5 more days of esomeprazole 40mg bid + levofloxacin 500mg bid + tinidazole 500 mg bid
  Interventions: Drug: Eradication therapy (amoxicillin; esomeprazole; tinidazole; levofloxacin)

INTERVENTIONS:
Drug: Eradication therapy (amoxicillin; esomeprazole; tinidazole; levofloxacin) — amoxicillin tablets 1 g; esomeprazole tablets 40mg; tinidazole tablets 500mg; levofloxacin tablets 500 mg
  Other Names: proton pump inhibitors

SUMMARY:
A five day quadruple concomitant therapy is as effective and safe as a 10 day sequential therapy for eradication of H. pylori infection.

DETAILED DESCRIPTION:
The investigators studied 180 consecutive patients with H. pylori infection who were randomized to 5-day concomitant therapy (90 patients) and to 10-day sequential therapy (90 patients). 6 and 10 weeks after the end of therapy, patients were evaluated for their H. pylori status by 13C Urea Breath Test. Side effects and costs of either regimen were evaluated. In patients whose H pylori status at entry was assessed by endoscopy, culture was performed and antimicrobial resistance was determined

ELIGIBILITY:
Inclusion Criteria:

* H. pylori-infected patients who were at least 18 years of age and who had never received H. pylori eradication treatment were included in the study.

Exclusion Criteria:

* previous treatment for H. pylori infection,
* use of inhibitors of acid secretion and/or antibiotics during the 6 weeks before the study,
* gastrointestinal malignancy,
* previous gastro-oesophageal surgery,
* severe concomitant cardiovascular,
* respiratory or endocrine diseases,
* clinically significant renal or hepatic disease,
* hematologic disorders,
* any other clinically significant medical condition that could increase risk,
* history of allergy to any of the drug used in the study,
* pregnancy or lactation,
* alcohol abuse,
* drug addiction,
* severe neurologic or psychiatric disorders, and
* long-term use of corticosteroids or anti-inflammatory drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Eradication Rate | 1 year
  The eradication rate obtained with the two treatments will be evaluated in the per-protocol and intention-to-treat analyses

SECONDARY OUTCOMES:
Adverse events | 1 year
  The incidence of adverse events during therapy will be assessed: bad taste, taste alteration, nausea, vomiting, diarrhoea, epigastric pain, glossitis, headache
Costs of either regimen | 1 year
  The costs related to each treatment will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Marco Romano, MD, Principal Investigator — Second University of Naples Medical School
Locations (1):
- Dipartimento di Internistica Clinica e Sperimentale, SUN, Naples, Napoli, Italy